CLINICAL TRIAL: NCT03677128
Title: A Mobile Health (mHealth) Case Management System for Reducing Pediatric Cancer Treatment Abandonment
Brief Title: Mobile Health Case Management System for Reducing Pediatric Treatment Abandonment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00094010; 1R21CA217268-01A1 (NIH)
Record Dates: First submitted 2018-08-21; First posted 2018-09-19 (Actual); Results first posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Burkitt Lymphoma; Retinoblastoma; Diffuse Large B-cell Lymphoma
Keywords: Digital Health; Pediatric Cancer; Low and middle-income country; Tanzania; Healthcare provider decision support; Protocol-driven treatment; Burkitt lymphoma; Retinoblastoma; Treatment abandonment; Client health records; Diffuse large B-cell lymphoma
MeSH Terms: conditions — Burkitt Lymphoma; Retinoblastoma; Lymphoma, Large B-Cell, Diffuse; Neoplasms

STUDY DESIGN:
Intervention Model Description: Effects on outcomes when using mNavigator will be compared to historical controls (preceding mNavigator use). Number of participants below references those who will be consented prospectively to participate in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mNavigator (Experimental): Allied health providers will use mNavigator to guide diagnosis and treatment for pediatric cancer patients at Bugando Medical Centre (BMC).
  Interventions: Other: mNavigator
- Historical controls (No Intervention): BL (DLBCL)/Rb retrospective patients (treated between 2015-2019) when standardized treatment protocols for BL (DLBCL) and Rb were introduced at BMC.

INTERVENTIONS:
Other: mNavigator — Allied health providers at BMC will use mNavigator to facilitate compliance with protocol-driven treatment and reduce patient abandonment for patients diagnosed with Burkitt lymphoma, Diffuse large B-cell lymphoma or retinoblastoma.
  Arms: mNavigator

SUMMARY:
Digital case management systems have the potential to increase compliance with protocol-driven treatment, reduce treatment abandonment and ultimately help to close the discrepancy in pediatric cancer outcomes between Low and Middle Income Countries (LMICs) and high-income countries (HICs). The investigators aim to adapt an open-source digital case management platform to incorporate standardized pediatric oncology protocols. Effectiveness will be evaluated by provider protocol compliance (primary outcome) and patient treatment abandonment rates using the digital case management system as compared to historic controls. The study population will include patients diagnosed with Burkitt lymphoma, Diffuse large B-cell lymphoma (DLBCL) or retinoblastoma at Bugando Medical Centre in Tanzania.

DETAILED DESCRIPTION:
Each year, approximately 220,000 children globally are newly diagnosed with cancer. Over 85% of these new diagnoses are made in low- and middle-income countries (LMICs). Survival rates in LMICs are 5-25% compared to 80% in high-income countries (HICs). One of the primary contributors to the discrepancy in survival outcomes between LMICs and HICs is a high rate of treatment abandonment, defined as refusal to initiate or failure to complete curative treatment. Treatment abandonment rate in Tanzania is higher than in other LMICs (40% compared to 10-25%), directly impacting patient survival. In HICs, protocol-driven treatment for children with cancer has led to increased treatment compliance and large improvements in survival. However, it is often not feasible or appropriate to use protocol-driven treatment in LMICs without necessary supportive care, human resources and infrastructure. Not surprisingly, protocol-related compliance is lower in LMICs compared to HICs. Digital technologies for health (i.e., digital health) can facilitate implementation of and compliance with standardized pediatric oncology protocols through step-by-step decision support algorithms, reminders and alerts related to patient visits, and timely data for health service coordination with allied health providers (e.g., nurses, pharmacists etc.). This multidisciplinary team from Duke University and Dimagi Inc. in USA, and Bugando Medical Centre (BMC) in Tanzania, proposes to adapt, implement, and evaluate a digital case management system, called mNavigator, at BMC to improve health provider compliance with standardized pediatric oncology protocols.

For Aim 1, mNavigator development will initially focus on the two nationally-approved protocols for Burkitt lymphoma and retinoblastoma. The treatment for Diffuse large B-cell lymphoma (DLBCL) follows the Burkitt lymphoma treatment protocol. Using principles of persuasive system design and the Consolidated Framework for Implementation Research (CFIR), prompts that guide users through protocol implementation will be used as behavioral triggers to assist with perceived ease of use.

For Aim 2, allied health providers at BMC will receive training on using mNavigator as part of an in-country workshop led by the M-PIs. This training will be followed by supported implementation. Following this training period, mNavigator will be used to enroll pediatric patients at BMC with pre-clinical diagnosis of BL, Diffuse large B-cell lymphoma (DLBCL) or Rb, over a period of over one and a half years and manage their care for the duration of treatment (up to 3 months for BL and DLBCL, and 4 months for Rb). BMC receives and treats approximately 150 patients every year, with an estimated 50 patients annually with Burkitt lymphoma (BL), Diffuse large B-cell lymphoma (DLBCL) or Rb. To review historic compliance, files of patients diagnosed after 2015 with BL, Diffuse large B-cell lymphoma (DLBCL) and Rb (when protocols were introduced) will be abstracted by trained research assistants. Compliance with protocol-driven treatment will be monitored using mNavigator. System functionality will be assessed. Semi-structured assessments of provider system acceptance and usability will be conducted along with elucidating caregiver reported barriers to treatment completion.

Secondary objective is to describe factors that facilitate or inhibit implementation of mNavigator.

ELIGIBILITY:
There are two categories of participants: Patients with Burkitt Lymphoma, Diffuse large B-cell lymphoma or retinoblastoma; and health providers at BMC who participate in testing and/or use of mNavigator. Eligibility criteria are as follows:

A) For patients:

*All patients will be registered in the pre-diagnosis cohort but, for the purposes of this study, primary and secondary outcomes will only be tracked for patients with BL, DLBCL or RB once the diagnosis is made.

Inclusion Criteria:

* Inclusion criteria are pediatric oncology patients diagnosed with Burkitt Lymphoma, Diffuse large B-cell lymphoma or Retinoblastoma under the age of 18

Exclusion criteria:

* Patients older than 18 years at registration
* Patients with diagnoses other than Burkitt lymphoma, Diffuse large B-cell lymphoma or retinoblastoma.

B) For providers:

Inclusion Criteria:

* Must be health provider or staff working at BMC who provides care for cancer patients.
* Must be 18 years of age or older.

Exclusion:

- Persons younger than 18 years of age.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Schroeder, MD MPH, Principal Investigator — Duke University; Lavanya Vasudevan, PhD, Principal Investigator — Duke University
Locations (1):
- Bugando Medical Centre, Mwanza, Lake Zone, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vasudevan L, Schroeder K, Raveendran Y, Goel K, Makarushka C, Masalu N, Zullig LL. Using digital health to facilitate compliance with standardized pediatric cancer treatment guidelines in Tanzania: protocol for an early-stage effectiveness-implementation hybrid study. BMC Cancer. 2020 Mar 29;20(1):254. doi: 10.1186/s12885-020-6611-3. PMID 32223740

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred July 2019 - April 2022. Due to COVID-19, in March 2020, the National Institute of Medical Research in Tanzania paused all clinical research activities in the country, stopping new enrollment until research activities resumed in August 2020.
Pre-assignment Details: Historical control patients were not considered enrolled, but historical control data was used as a comparison, so is included here. mNavigator users were also not considered enrolled, but provided data.
Groups:
- mNavigator - Burkitt Lymphoma (BL): Prospective cohort of patients diagnosed with BL where allied health providers used mNavigator to guide diagnosis and treatment at Bugando Medical Centre (BMC).
  mNavigator: Allied health providers at BMC will use mNavigator to facilitate compliance with protocol-driven treatment and reduce patient abandonment for patients diagnosed with Burkitt lymphoma, Diffuse large B-cell lymphoma (DLBCL) or retinoblastoma.
- mNavigator - Retinoblastoma (Rb): Prospective cohort of patients diagnosed with Rb where allied health providers used mNavigator to guide diagnosis and treatment at Bugando Medical Centre (BMC).
  mNavigator: Allied health providers at BMC will use mNavigator to facilitate compliance with protocol-driven treatment and reduce patient abandonment for patients diagnosed with Burkitt lymphoma, Diffuse large B-cell lymphoma (DLBCL) or retinoblastoma.
- Historical Controls - Burkitt Lymphoma (BL): BL retrospective patients (treated between 2015-2019) when standardized treatment protocols for BL (DLBCL) and Rb were introduced at Bugando Medical Centre (BMC).
- Historical Controls - Retinoblastoma (Rb): Rb retrospective patients (treated between 2015-2019) when standardized treatment protocols for BL (DLBCL) and Rb were introduced at Bugando Medical Centre (BMC).
- mNavigator Users: Health care providers using mNavigator
Period: Overall Study
Arm/Group | mNavigator - Burkitt Lymphoma (BL) | mNavigator - Retinoblastoma (Rb) | Historical Controls - Burkitt Lymphoma (BL) | Historical Controls - Retinoblastoma (Rb) | mNavigator Users
Started | 46 | 29 | 63 | 25 | 4
Completed | 36 | 16 | 63 | 25 | 4
Not Completed | 10 | 13 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who completed the study. Baseline Characteristics not collected on mNavigator Users.
Groups:
- Total: Total of all reporting groups
Arm/Group | mNavigator - Burkitt Lymphoma (BL) | mNavigator - Retinoblastoma (Rb) | Historical Controls - Burkitt Lymphoma (BL) | Historical Controls - Retinoblastoma (Rb) | mNavigator Users | Total
Number analyzed (Participants) | 36 | 16 | 63 | 25 | 0 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.2 (4.3) | 2.8 (1.6) | 9.5 (4.0) | 3.3 (1.6) |  | 5.95 (3.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 27 | 12 |  | 55
  Male | 27 | 9 | 36 | 13 |  | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 |  | 0
  Not Hispanic or Latino | 36 | 16 | 63 | 25 |  | 140
  Unknown or Not Reported | 0 | 0 | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 |  | 0
  Asian | 0 | 0 | 0 | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 |  | 0
  Black or African American | 36 | 16 | 63 | 25 |  | 140
  White | 0 | 0 | 0 | 0 |  | 0
  More than one race | 0 | 0 | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Tanzania | 36 | 16 | 63 | 25 |  | 140

OUTCOME MEASURES:

1. Primary Outcome: Protocol Compliance as Measured by Percent Compliance to Prescribed Chemotherapy
Time Frame: Approximately 1 year
Population: Participants who completed the study and historical controls. Does not apply to mNavigator Users.
Measure: Mean (Standard Deviation); unit: percentage of compliance
Arm/Group | mNavigator - Burkitt Lymphoma (BL) | mNavigator - Retinoblastoma (Rb) | Historical Controls - Burkitt Lymphoma (BL) | Historical Controls - Retinoblastoma (Rb) | mNavigator Users
Number analyzed (Participants) | 36 | 16 | 63 | 25 | 0
percentage of compliance | 73.8 (15.1) | 96.0 (5.1) | 50.0 (16.0) | 74.9 (11.9) |
Statistical Analysis 1: Comparison: mNavigator - Burkitt Lymphoma (BL) vs Historical Controls - Burkitt Lymphoma (BL); Test type: Other; p < 0.001, Kruskal-Wallis; Mean Difference (Final Values) = 23.8
Statistical Analysis 2: Comparison: mNavigator - Retinoblastoma (Rb) vs Historical Controls - Retinoblastoma (Rb); Test type: Other; p < 0.001, Kruskal-Wallis; Mean Difference (Final Values) = 21.1

2. Secondary Outcome: Time to Diagnosis (in Days)
Description: The number of days to diagnosis using mNavigator compared to historical controls. Time to diagnosis is computed as the duration (in days) from registration at oncology clinic to confirmatory diagnosis. If diagnosis was determined prior to intake, 0 days was entered.
Time Frame: Approximately 1 year
Population: Participants who completed the study and historical controls. Does not apply to mNavigator Users.
Measure: Median (Standard Deviation); unit: days
Arm/Group | mNavigator - Burkitt Lymphoma (BL) | mNavigator - Retinoblastoma (Rb) | Historical Controls - Burkitt Lymphoma (BL) | Historical Controls - Retinoblastoma (Rb) | mNavigator Users
Number analyzed (Participants) | 36 | 16 | 63 | 25 | 0
days | 0 (3.3) | 0 (0.5) | 5 (145.9) | 0 (1.0) |

3. Secondary Outcome: Number of Participants Who Abandon Treatment
Description: Treatment abandonment is defined as missing 4 or more consecutive weeks of treatment or follow-up while on therapy.
Time Frame: Approximately 1 year
Population: Participants who completed the study and historical controls. Does not apply to mNavigator Users.
Measure: Count of Participants; unit: Participants
Arm/Group | mNavigator - Burkitt Lymphoma (BL) | mNavigator - Retinoblastoma (Rb) | Historical Controls - Burkitt Lymphoma (BL) | Historical Controls - Retinoblastoma (Rb) | mNavigator Users
Number analyzed (Participants) | 36 | 16 | 63 | 25 | 0
Participants | 9 | 5 | 25 | 18 |

4. Secondary Outcome: Number of Participants Who Completed Treatment as Indicated
Description: Patients registered in mNavigator who completed treatment as indicated (excludes patient deaths or abandoned care without returning, treatment failure, and Rb patients who should have enucleation per protocol but did not complete).
Time Frame: Approximately 1 year after treatment initiation
Population: Participants who completed the study and historical controls. Does not apply to mNavigator Users.
Measure: Count of Participants; unit: Participants
Arm/Group | mNavigator - Burkitt Lymphoma (BL) | mNavigator - Retinoblastoma (Rb) | Historical Controls - Burkitt Lymphoma (BL) | Historical Controls - Retinoblastoma (Rb) | mNavigator Users
Number analyzed (Participants) | 36 | 16 | 63 | 25 | 0
Participants | 23 | 10 | 25 | 3 |

5. Other Pre Specified Outcome: System Usability Scale Score
Description: System usability scale (SUS) score ranging from 0-100 measured using a 10-point validated system usability scale. A SUS score above 68 is considered above average usability.
Time Frame: Approximately 1 year
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Monthly Utilization of mNavigator
Description: Number of forms submitted using mNavigator, stratified, by users, per month of implementation.
Time Frame: Approximately 1 year
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Number of Instances of mNavigator Failure Per Month (All-causes)
Time Frame: Approximately 1 year
Population: Only applies to mNavigator Users.
Measure: Mean (Standard Deviation); unit: failures per month
Arm/Group | mNavigator Users
Number analyzed (Participants) | 4
failures per month | 0 (0)

8. Other Pre Specified Outcome: Number of Instances of CommCare Failure Per Month (All-causes)
Description: Number of instances of CommCare failure per month (all-causes)
Time Frame: Approximately 1 year
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Number of Instances of Device Failure Per Month (All-causes)
Description: Number of instances of device failure per month (all-causes)
Time Frame: Approximately 1 year
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Number of Hours of Initial Training as Well as Hours of Ongoing Support Provided During the First Month of Implementation
Description: Number of hours of initial training as well as hours of ongoing support provided during the first month of implementation
Time Frame: Approximately 1 year
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Number of Users Who Are Proficient in Use of mNavigator Within First Month of Implementation
Description: Number of users who are proficient in use of mNavigator within first month of implementation
Time Frame: Approximately 1 year
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Average Time in Minutes Spent Completing Each Form, Stratified by Form
Description: Average time in minutes spent completing each form, stratified by form
Time Frame: Approximately 1 year
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Time Per Patient
Description: Total time in minutes spent entering patient data in mNavigator, from time of registration until an outcome is recorded. Calculated by summing time for completing each form, by patient.
Time Frame: Approximately 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Approximately 1 year from treatment initiation
Description: Adverse Event data not collected on historical controls or mNavigator users.
Arm/Group | mNavigator - Burkitt Lymphoma (BL) | mNavigator - Retinoblastoma (Rb) | Historical Controls - Burkitt Lymphoma (BL) | Historical Controls - Retinoblastoma (Rb) | mNavigator Users
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/29 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/29 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/46 | 0/29 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/28/NCT03677128/Prot_SAP_000.pdf